CLINICAL TRIAL: NCT05040152
Title: Address Obesity to Reduce Cancer Risk and Health Disparities in Rural Ohio
Brief Title: Weight Loss Intervention for the Reduction of Cancer Risk and Health Disparities in Rural Ohio
Acronym: HERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-21007; NCI-2021-03973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); F99CA253745 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-09-10 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (telephone-based intervention) (Experimental): Participants receive weekly telephone-based weight loss intervention for 15 weeks, including dietary recommendations tailored to their current weight and weight loss target, home-based aerobic and resistance exercise, and weekly telephone counseling session over 30-45 minutes.
  Interventions: Behavioral: Dietary Counseling and Surveillance; Other: Exercise Intervention; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention
- Arm II (education brochures) (Active Comparator): Participants receive education brochures describing the American Institute for Cancer Research physical activity and dietary guidelines.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Dietary Counseling and Surveillance — Receive dietary recommendations
  Arms: Arm I (telephone-based intervention)
Other: Exercise Intervention — Complete home exercises
  Arms: Arm I (telephone-based intervention)
Other: Informational Intervention — Receive education brochures
  Arms: Arm II (education brochures)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone-based weight loss intervention
  Arms: Arm I (telephone-based intervention)

SUMMARY:
This study determines the feasibility of a telephone-based weight lost intervention in reducing cancer risk and health disparities in rural Ohio. Obesity is the leading preventable cause of cancer, and obesity-related inflammation is linked to elevated cancer risk, independent of obesity itself. Rural populations are a vulnerable population in need of increased access to tailored strategies and benefit from weight loss interventions. This study aims to see whether a telephone-based intervention may help obese people in rural area to reduce body weight, so as to prevent obesity-related cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and acceptability of a 15-week telephone-based weight loss intervention among overweight/obese rural residents.

II. To estimate the preliminary efficacy of the lifestyle modifications on weight loss, body composition (fat mass, percent body fat), inflammatory biomarkers (IL-6, TNF-alpha, and C-recreative protein [CRP]), and other disease risk factors (lipid profiles).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive weekly telephone-based weight loss intervention for 15 weeks, including dietary recommendations tailored to their current weight and weight loss target, home-based aerobic and resistance exercise, and weekly telephone counseling session over 30-45 minutes.

ARM II: Participants receive education brochures describing the American Institute for Cancer Research physical activity and dietary guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >= 25 kg/m^2
* Age: 20-64.9 years
* Not currently participating in any weight loss intervention or meet the physical activity recommendation (150 min/week of moderate-intensity exercise or 75 min/week of vigorous exercise)
* The ability to walk two blocks
* Ability to speak and read English

Exclusion Criteria:

* Prior cancer diagnosis (except non-melanoma skin cancer) or severe medical conditions such as unstable cardiovascular disease or digestive disorders that would preclude physical activity and dietary intervention
* Pregnant or nursing women
* Unable to give informed consent

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Focht, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures)
Started | 27 | 13
Completed | 22 | 11
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures) | Total
Number analyzed (Participants) | 27 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 13 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 13 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 13 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a 15-week Telephone-based Weight Loss Intervention
Description: Will be defined as the number of enrolled participants who complete the study.
Time Frame: Up to 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures)
Number analyzed (Participants) | 27 | 13
Participants | 22 | 11

2. Secondary Outcome: Changes in Body Weight (KG)
Description: Changes in body weight (KG)will be measured by a weight scale
Time Frame: Up to 15 weeks
Population: The number of participants analyzed is the number that the 15 week intervention and the 15 week follow-up
Measure: Mean (Standard Error); unit: kg
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures)
Number analyzed (Participants) | 22 | 11
kg | -4.93 (1.12) | -2.09 (1.58)

3. Secondary Outcome: Changes in Body Fat Mass
Description: Changes in body fat mass will be measured using a 3-Dimension (3D) Body Scanner, Styku S100
Time Frame: Up to 15 weeks
Measure: Mean (Standard Error); unit: lb
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures)
Number analyzed (Participants) | 22 | 11
lb | 0.23 (3.46) | 0.11 (2.38)

4. Other Pre Specified Outcome: Changes Body Fat Percentage
Description: Changes body fat percentage will be measured using a 3-Dimension (3D) Body Scanner, Styku S100
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Lipid Profiles
Description: Total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), and low-density lipoprotein cholesterol (LDL-C) will be obtained by fasting capillary blood sampling from fingerstick and analyzed using Cholestech LDX
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: C-reactive Protein (CRP) Concentration (ng/L)
Description: C-reactive protein (CRP) concentration (ng/L) will be quantified with an automated chemistry analyzer
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Interleukin (IL)-6 Concentration (pg/mL)
Description: Interleukin (IL)-6 concentration (pg/mL) will be quantified with sandwich enzyme immunoassay assays
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: TNF-alpha Concentration (pg/mL)
Description: TNF-alpha concentration (pg/mL) will be quantified with sandwich enzyme
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Physical Fitness
Description: Participants will be asked to complete two valid and reliable timed performance-related mobility tasks, including 400-meter walk and lift and carry task
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Physical Activity
Description: Self-reported using Leisure-Time Exercise Questionnaires118. Objectively measured physical activity will be recorded using the LIFECORDER Plus Accelerometer for 7 days in the 1st and 15th week
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exercise-Related Self-Efficacy Exercise-Related
Description: Assessed by using Exercise Self-Efficacy, Barrier Self-Efficacy, and Multi-dimensional Self-Efficacy scales
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Dietary Intake
Description: Self-reported using the National Institutes of Health Daily Food List
Time Frame: Up to 15 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 15 weeks
Arm/Group | Arm I (Telephone-based Intervention) | Arm II (Education Brochures)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 0/27 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05040152/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT05040152/ICF_001.pdf